CLINICAL TRIAL: NCT00800137
Title: Bridge or Continue Coumadin for Device Surgery Randomized Controlled Trial (BRUISE CONTROL)
Brief Title: Bridge or Continue Coumadin for Device Surgery Randomized Controlled Trial
Acronym: BRUISECONTROL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: At time of pre-specified 2nd interim analysis
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, David Birnie, MD, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOHI-02
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Hematoma
Keywords: coumadin; device surgery; pocket hematoma; Pocket hematoma and device surgery
MeSH Terms: conditions — Hematoma | interventions — Heparin, Low-Molecular-Weight; Heparin; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bridging anti-coagulation (Active Comparator): Low Molecular Weight Heparin or IV unfractionated Heparin
  Interventions: Drug: low molecular weight heparin or unfractionated heparin
- Continued oral anti-coagulation (Experimental): Coumadin
  Interventions: Drug: Warfarin or coumadin

INTERVENTIONS:
Drug: low molecular weight heparin or unfractionated heparin — For elective patients with greater than 5 days pre-implant; discontinue oral anti-coagulation (coumadin) 5 days before the procedure. Full therapeutic doses of subcutaneous LMWH 3 days before the procedure.
  Patients with less than 5 days to implant can be given vitamin K (up to 2 mg) at the investigator discretion and start full therapeutic doses of either subcutaneous LMWH or IV Unfractionated Heparin (choice is at investigator's discretion) when INR is below the upper limit of the prescribed therapeutic range for the patient (usually greater than or equal to 2; 2.5 for some valve patients) and surgery to proceed when INR is less than 1.6.
  Last dose given in the morning(ie. > 24 hours)of the day prior to the procedure.
  Oral anti-coagulation (coumadin) will be resumed on the evening of the procedure.
  Full dose LMWH or full dose IV heparin will be restarted 24 hours after surgery.
  Arms: Bridging anti-coagulation
Drug: Warfarin or coumadin — Continue on oral anti-coagulant (coumadin). INR on the day of surgery will be < 3.0
  Arms: Continued oral anti-coagulation

SUMMARY:
Many cardiac patients requiring device (defibrillator or pacemaker) related surgery are on chronic oral anticoagulation therapy (usually coumadin). The risk of blood clot formation related to stopping oral anti-coagulant therapy is currently managed by using bridging heparin therapy in patients with moderate to high risk of blood clot formation. There is a substantial risk of bleeding in the pocket where the device is situated (pocket hematoma)related to bridging therapy. The purpose of this study is to compare the current standard of care of bridging with heparin to an experimental strategy of continuing coumadin therapy in higher risk patients undergoing device surgery, with the hypothesis being that the continued oral anti-coagulation group will have a lower pocket hematoma rate as compared to the bridging with heparin group.

DETAILED DESCRIPTION:
Eligible patients will be equally randomized (1:1) to the Conventional/control arm (bridging anti-coagulation)or to the Experimental arm (continued coumadin). In the Conventional arm there are 2 options. Patients with greater than 5 days pre-implant will discontinue oral anti-coagulant (coumadin) 5 days before the procedure,and start full therapeutic doses of subcutaneous low molecular weight heparin (LMWH)3 days before the procedure. Patients with less than 5 days to implant can be given Vitamin K at the investigator's discretion and start full therapeutic doses of either subcutaneous LMWH or IV unfractionated Heparin (choice is at investigator discretion) when the INR is below the therapeutic range for the patient (usually greater than or equal to 2; 2.5 for some valve patients) and surgery to proceed when INR is less than 1.6. Oral anti-coagulant (coumadin) will resume on the evening of the procedure. Full dose LMWH injections or full dose IV heparin will be started 24 hours after surgery.

In the Experimental arm patients will continue on their oral anti-coagulant (coumadin). The INR on the day of surgery will be < 3.0.

ASA will be continued in all patients. Plavix will be continued in patients with drug-eluting stents.

Patients will be monitored for the development of any hematoma or bleeding event during admission. There will be a unblinded team responsible for device implant and follow-up and a blinded team responsible to monitor any bleeding events or hematoma and determine if it meets the primary endpoint criteria for the study. The blinded team will have no knowledge of the treatment arm and will be involved only if the patient develops a hematoma or bleeding event. All hematomas and bleeding events will be followed until resolution.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient undergoing elective device surgery (i.e. de novo device implantation or pulse generator change or lead replacement or pocket revision)
2. Patient at moderate or high risk of arterial thrombo-embolic events (ATE) or high risk of venous thrombo-embolic events (VTE) (defined as one or more of following):

   * Prosthetic mitral valve replacement
   * Caged ball or tilting disc aortic valve prosthesis
   * Bileaflet aortic valve prosthesis and one or more of: AF (atrial Fibrillation/Atrial Flutter), prior stroke or TIA, hypertension, diabetes, CHF age >75
   * AFib/Flutter associated with rheumatic valvular heart disease
   * Non-rheumatic AFib/Flutter and CHADS2 risk criteria SCORE > 2
   * Non-rheumatic AFib/Flutter and stroke or TIA (within 3 months)
   * Persistent/permanent AFib/Flutter on day of acceptance for device surgery AND plan for cardioversion or DFT testing at device implant
   * Recent (within 3 months) VTE
   * Severe thrombophilia (Protein C or S deficiency or anti-thrombin or anti-phospholipid antibodies or multiple abnormalities)
3. Willing to self-inject or have a relative or friend or nurse inject LMWH

Exclusion Criteria:

1. Unable ro unwilling to provide informed consent
2. History of noncompliance of medical therapy
3. Renal failure with Cr > 180 umol/l
4. Prior Heparin induced thrombocytopenia
5. Active device infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2008-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Clinically significant hematoma (defined as hematoma requiring reoperation and/or transfusion and/or unplanned or prolonged hospitalization and/or interruption of LMWH or IV heparin or oral anti-coagulant. | Device implant until first routine post-op visit

SECONDARY OUTCOMES:
Components of the primary outcome,composite of all other major peri-operative bleeding events and thrombo-embolic events. | Device implant to first routine post-op visit

CONTACTS AND LOCATIONS:
Overall Officials: David Birnie, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (22):
- Instituto de Cardiologia - Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (21):
  - University of Calgary, Calgary, Alberta
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - St. John Regional Hospital, Saint John, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Science Center, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Sciences Center, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Rouge Valley Hospital, Scarborough Village, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Mike's Hospital, Toronto, Ontario
  - Cité-de-la-Santé Hospital, Laval, Quebec
  - Centre Hospitalier de L'Université de Montréal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Hôpital Sacré-Coeur de Montréal, Montreal, Quebec
  - Hôpital Laval, Québec, Quebec
  - Sherbrooke University Hospital Centre CHUS, Sherbrooke, Quebec

REFERENCES:
- [Result] Birnie DH, Healey JS, Wells GA, Verma A, Tang AS, Krahn AD, Simpson CS, Ayala-Paredes F, Coutu B, Leiria TL, Essebag V; BRUISE CONTROL Investigators. Pacemaker or defibrillator surgery without interruption of anticoagulation. N Engl J Med. 2013 May 30;368(22):2084-93. doi: 10.1056/NEJMoa1302946. Epub 2013 May 9. PMID 23659733
- [Derived] Essebag V, Healey JS, Joza J, Nery PB, Kalfon E, Leiria TLL, Verma A, Ayala-Paredes F, Coutu B, Sumner GL, Becker G, Philippon F, Eikelboom J, Sandhu RK, Sapp J, Leather R, Yung D, Thibault B, Simpson CS, Ahmad K, Toal S, Sturmer M, Kavanagh K, Crystal E, Wells GA, Krahn AD, Birnie DH. Effect of Direct Oral Anticoagulants, Warfarin, and Antiplatelet Agents on Risk of Device Pocket Hematoma: Combined Analysis of BRUISE CONTROL 1 and 2. Circ Arrhythm Electrophysiol. 2019 Oct;12(10):e007545. doi: 10.1161/CIRCEP.119.007545. Epub 2019 Oct 15. PMID 31610718
- [Derived] Essebag V, AlTurki A, Proietti R, Healey JS, Wells GA, Verma A, Krahn AD, Simpson CS, Ayala-Paredes F, Coutu B, Leather R, Ahmad K, Toal S, Sapp J, Sturmer M, Kavanagh K, Crystal E, Leiria TLL, Seifer C, Rinne C, Birnie D; BRUISE CONTROL Investigators. Concomitant anti-platelet therapy in warfarin-treated patients undergoing cardiac rhythm device implantation: A secondary analysis of the BRUISE CONTROL trial. Int J Cardiol. 2019 Aug 1;288:87-93. doi: 10.1016/j.ijcard.2019.04.066. Epub 2019 Apr 26. PMID 31056413
- [Derived] Essebag V, Verma A, Healey JS, Krahn AD, Kalfon E, Coutu B, Ayala-Paredes F, Tang AS, Sapp J, Sturmer M, Keren A, Wells GA, Birnie DH; BRUISE CONTROL Investigators. Clinically Significant Pocket Hematoma Increases Long-Term Risk of Device Infection: BRUISE CONTROL INFECTION Study. J Am Coll Cardiol. 2016 Mar 22;67(11):1300-8. doi: 10.1016/j.jacc.2016.01.009. PMID 26988951